CLINICAL TRIAL: NCT06370078
Title: Effect of Early Administration of Albumin 20% Versus Crystalloid During Resuscitation of Patient With Septic Shock: a Randomized Controlled Trial
Brief Title: Effect of Early Administration of Albumin 20% Versus Crystalloid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ahmed Helal
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Serum Albumin, Human; Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Albumin Group (Experimental): About 23 patients will be objected for resuscitation with 60 gm (300 ml) human albumin 20% (HA 20%) over 2-3 hours combined usual practice with 30 ml/kg crystalloid.
  Interventions: Drug: Albumin Human
- Control Group (Active Comparator): About 23 patients will be objected for resuscitation with 30 ml/kg crystalloid.
  Interventions: Drug: Albumin Human

INTERVENTIONS:
Drug: Albumin Human — To investigate the effect of early administration of albumin in the ICU after onset of septic shock compared to volume replacement therapy without albumin on patient outcome.
  Other Names: crystalloids

SUMMARY:
Sepsis and septic shock are global health problems, leading to a high mortality rate. They are often associated with extremely low blood pressure and multiple organ dysfunctions, which are the main causes of death in critically ill patients. Fluid resuscitation is one of the most critical treatments for patients with sepsis and septic shock.

An early administration of an appropriate fluid to patients is considered the most effective way to increase blood pressure, improve tissue perfusion, and save their lives. Crystalloid fluids are a subset of intravenous solutions composed of mineral salts and other small, water-soluble molecules, including normal, isotonic or hypertonic saline, and various buffered solutions.

DETAILED DESCRIPTION:
Crystalloid fluids are a subset of intravenous solutions composed of mineral salts and other small, water-soluble molecules, including normal, isotonic or hypertonic saline, and various buffered solutions.

Colloid solutions are composed of various amounts of substances, for instance, albumin, hydroxyethyl starch, dextran, and gelatine. Although the current international guidelines from the Surviving Sepsis Campaign recommend crystalloids to perform the initial resuscitation, and the replacement with albumin on patients who require substantial amounts of crystalloids, the choice of the best type of resuscitation fluids is still under debate.

Albumin, in addition to its oncotic functions, has a variety of other properties, including binding and transport of various endogenous molecules, anti-inflammatory and anti-oxidative effects, and modulation of nitric oxide metabolism.These properties are particularly relevant in critically ill patients, especially in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of septic shock that meets all the following Criteria: Clinically possible, probable, or microbiologically confirmed infection according to the definitions of the International-Sepsis- Forums (ISF), Despite adequate volume therapy, vasopressors are required to maintain mean arterial pressure (MAP) ≥ 65 mmHg for at least 1 hour, Serum lactate concentration > 2 mmol/l (18 mg/dl) despite adequate volume therapy.
* Onset of septic shock less than 24 h prior to study inclusion.
* Women of childbearing age: negative pregnancy test

Exclusion Criteria:

* Moribund conditions
* End of life decisions
* Previous participation to this trial or any other interventional clinical trial
* Known hypersensitivity to albumin or any component of the trial drug
* Clinical conditions, where albumin administration may be unfavourable
* Breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Recovery from shock | 3 Hours
  A reversal of hypotension (MAP) at the end of the first three hours of the resuscitation period.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmed Mohamed, Professor, Study Chair — ICU department , Faculty of Medicine, Assuit University
Locations (1):
- Assuit University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided